CLINICAL TRIAL: NCT05622487
Title: The Effects of Neural Therapy and Kinesio Taping on Pain, Functional Status, and Quality of Life in Fibromyalgia Patients: A Prospective Randomized Double-Blind Study
Brief Title: Neural Therapy and Kinesio Taping Effectiveness in Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Sinan GOK, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Istanbul Universty FMS
Record Dates: First submitted 2022-08-06; First posted 2022-11-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Neural Therapy; Kinesio Taping
MeSH Terms: conditions — Fibromyalgia | interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neural Therapy (Active Comparator): Segmental neural therapy will be administered with intradermal 0.5% lidocaine from cervical 1st to sacral 1st vertebra and upper trapezius region with quaddel injections.. Sham kinesio taping will be applied to the bilateral arms of the patients. Home exercise program; trapezius stretching, cervical, thoracic and lumbar paravertebral muscle stretching exercises will be required to be performed 10 times and every day.
  Interventions: Other: Neural Therapy
- Kinesio Taping (Active Comparator): Kinesio taping will be applied with muscle inhibition technique by stretching from the origin to the insertion of the upper trapezius, cervical thoracic and lumbar paravertebral muscles. Sham neural therapy will be applied to the bilateral arms of the patients. Home exercise program; trapezius stretching, cervical, thoracic and lumbar paravertebral muscle stretching exercises will be required to be performed 10 times and every day.
  Interventions: Other: Kinesio taping

INTERVENTIONS:
Other: Neural Therapy — Neural therapy is a form of treatment that aims to act on the autonomic nervous system, by injecting local anesthetics into certain parts of the body.
  Arms: Neural Therapy
Other: Kinesio taping — Kinesiotape is used for injury prevention, rehabilitation and performance enhancement. It has been shown to be clinically effective in increasing joint movements, increasing muscle activity, inducing muscle maximum torque earlier, and improving functional performance
  Arms: Kinesio Taping

SUMMARY:
The aim of this study; to investigate the effects of neural therapy and kinesio taping treatments on pain, functional status and quality of life in women with fibromyalgia.

DETAILED DESCRIPTION:
Fibromyalgia is a chronic disorder characterized by widespread pain, fatigue, sleep disturbance, cognitive impairment, and other physical symptoms that negatively affect physical and sensory functions and impair quality of life. Neural therapy and kinesio taping are treatments for musculoskeletal diseases. In this prospective, randomized controlled, double-blind, interventional study, 64 patients aged 18-55 years who met the eligibility criteria will be included in the study. Eligible participants will be randomly assigned to one of two groups using computer generated random numbers. Segmental neural therapy and sham kinesio taping will be applied to the first group. In the second group, kinesio taping with inhibition technique will be applied to bilateral trapezius and erector spina muscles and sham neural therapy will be added. Treatments will be applied once a week for a total of 6 weeks. Both groups will be given a home exercise program consisting of stretching exercises and will be checked every week. During the follow-up period, patients will be asked not to make changes to their current medical treatment. Participants will be evaluated for pain by Visual Analogue Scale (VAS), Fibromyalgia Impact Questionnaire (FIQ), Central Sensitisation Inventory (CSI), Beck Depression Inventory (BDI), Beck Anxiety Inventory (BAI), Health Assessment Questionnaire (HAQ), Short Form-36 (SF-36), manual algometer measurements and number of tender points, as well as post-treatment and post-treatment 3 month control data.

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed with fibromyalgia according to the ACR 2016 diagnostic criteria.
* Being a woman between the ages of 18 and 55.
* No change in the medical treatment he received for fibromyalgia syndrome during the study
* To be able to come to treatment 1 day a week for 6 weeks

Exclusion Criteria:

* Presence of known central nervous system or peripheral nervous system disease, progressive neurological deficit
* Peripheral venous insufficiency, coagulopathies and anticoagulant drug use
* Loss of sensation, loss of position sense, unhealed fracture or open surgical wound
* Uncontrolled hypertension and uncontrolled diabetes
* Be in major depression
* Cognitive impairment that causes difficulty following simple commands
* Pregnancy
* Be in menopause
* Allergy to local anesthetics and kinesio taping
* Open wound or infection at the application site

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale pain (0-10 point). | up to 3 month
  Higher scores mean a worse outcome
Fibromyalgia Impact Questionnaire (0-100 point) | up to 3 month
  The Fibromyalgia Impact Questionnaire was developed to assess the current functional status of women with FMS. Higher scores mean a worse outcome
Pain measurement with manual algometer | up to 3 month
  18 tender points in 1990 ACR FMS criteria will be evaluated with a manual algometer. Higher scores mean a worse outcome

SECONDARY OUTCOMES:
Beck Depression Inventory (0-63 point) | up to 3 month
  Beck Depression Inventory (BDI) is a frequently used evaluation criterion as a diagnosis and follow-up parameter in evaluating the state of depression. Higher scores mean a worse outcome
Beck Anxiety Inventory (0-63 point) | up to 3 month
  The scale aims to determine the frequency and severity of anxiety symptoms experienced by individuals. The highest score that can be obtained from the 21-item scale is 63. Higher scores mean a worse outcome
Central Sensitisation Inventory (0-100 point) | up to 3 month
  Central sensitization scale; It is a scale used to detect central sensitization conditions such as fibromyalgia, migraine, myofascial pain, temporomandibular disorder. Higher scores mean a worse outcome
Health Assessment Questionnaire (0-60 point) | up to 3 month
  The health assessment questionnaire shows the extent of the participant's functional ability, is sensitive to change, and is a good predictor of future cost and disability. Higher scores mean a worse outcome
Short Form-36 (0-100 point) | up to 3 month
  Short Form-36 is one of the commonly used scales in which health concepts such as functional status and well-being are evaluated. This scale examines health in 8 dimensions: physical function, physical role limitations, emotional role limitations, social function, mental health, vitality (energy), pain and general perception of health. Higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ayşegül Ketenci, Professor, Principal Investigator — Study Director
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul University Istanbul Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Istanbul, Fatıh
  - Istanbul University, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided